CLINICAL TRIAL: NCT03554616
Title: Efficacy of Three Different Bi-treated Long Lasting Insecticidal Nets and Deployment Strategy for Control of Malaria Transmitted by Pyrethroid Resistant Vectors: A Randomised Controlled Trial
Brief Title: Efficacy of Three Novel Bi-treated Long Lasting Insecticidal Nets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Kilimanjaro Christian Medical Centre, Tanzania (Other); National Institute for Medical Research, Tanzania (Other Government); University of Ottawa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ITDCZN11
Record Dates: First submitted 2018-04-26; First posted 2018-06-13 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2022-04

CONDITIONS: Malaria; Anaemia
Keywords: Malaria; Vector Control; Long lasting Insecticidal Net
MeSH Terms: conditions — Malaria; Anemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pyriproxyfen LLIN (Experimental): Royal Guard® (Disease Control Technologies, LLC) is a Long Lasting Insecticidal Net made of polyethylene incorporating a mixture of 225 mg/m2 pyriproxyfen and 261mg/m2 alpha-cypermethrin. This LLIN will be distributed to all the households in 21 clusters on a 1 LLIN per two household residents basis.
  Interventions: Other: pyriproxyfen LLIN
- Chlorfenapyr LLIN (Experimental): Interceptor® G2 (BASF corporation) is a LLIN made of polyester coated with a wash-resistant formulation of 200 mg/m2 chlorfenapyr and 100 mg/m2 alpha-cypermethrin. This LLIN will be distributed to all the households in 21 clusters on a 1 LLIN per two household residents basis.
  Interventions: Other: Chlorfenapyr LLIN
- Piperonyl butoxide LLIN (Experimental): Olyset® Plus (Sumitomo Chemicals) is a LLIN combining Piperonyl butoxide (400mg/m2) and the repellent pyrethroid permethrin (800 mg/m2) incorporated into the polyethylene fibres. This LLIN will be distributed to all the households in 21 clusters on a 1 LLIN per two household residents basis.
  Interventions: Other: Piperonyl butoxide LLIN
- Standard LLIN (Active Comparator): Interceptor® (BASF Corporation) is a single pyrethroid-treated LLIN with alpha-cypermethrin (coated onto filaments) at a target dose of 200 mg/m2 of polyester fabric. This LLIN will be distributed to all the households in 21 clusters on a 1 LLIN per two household residents basis.
  Interventions: Other: Standard LLIN

INTERVENTIONS:
Other: Chlorfenapyr LLIN — Dual active ingredient Long Lasting Insecticidal Net
  Arms: Chlorfenapyr LLIN
Other: pyriproxyfen LLIN — Dual active ingredient Long Lasting Insecticidal Net
  Arms: Pyriproxyfen LLIN
Other: Piperonyl butoxide LLIN — Combination insecticide and synergist Long Lasting Insecticidal Net
  Arms: Piperonyl butoxide LLIN
Other: Standard LLIN — Standard Long Lasting Insecticidal Net with one insecticide
  Arms: Standard LLIN

SUMMARY:
The massive scale-up of Long Lasting Insecticidal Nets (LLIN) has led to a major reduction in malaria burden (up to 50%) in many sub-Saharan African countries. This progress is threatened by the wide scale selection of insecticide resistant malaria vectors. New types of LLIN combining a mixture of two insecticides or an insecticide and a synergist have been developed to control resistant mosquitoes.

The efficacy of three bi-treated LLIN are compared to a standard LLIN in a four-arm, single blinded, cluster-randomized trial in Misungwi district, Tanzania. The arms are; 1/ Royal Guard, a net combining pyriproxyfen (PPF), which is known to disrupt female reproduction and fertility of eggs, and the pyrethroid alpha-cypermethrin, 2/Interceptor G2, LLIN incorporating a mixture of two adulticides with different modes of action; chlorfenapyr and a pyrethroid (alpha-cypermethrin), and 3/ Olyset Plus an LLIN which incorporates a synergist, piperonyl butoxide (PBO), to enhance the potency of pyrethroid insecticides, and 4/ The control arm: Interceptor treated a standard LLIN treated with alpha-cypermethrin.

The primary outcome of the trial will be cross-sectional community prevalence of malaria infection (by RDT) in children aged 6 months to 14 years at 12 and 24 months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* At least one child between 6 months to 14 years old having permanent residence in selected household
* Having an adult caregiver willing to provide written consent for the household and clinical survey

Exclusion Criteria:

* Dwelling not found or vacant during the survey
* No adult caregiver capable to give informed consent
* Children severely ill

Ages: 6 Months to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4200 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Malaria infection prevalence in children 6 months to 14 years | 24 months post intervention
  Malaria prevalence will be assessed using Malaria Rapid Diagnostic test (CareStart Malaria histidine-rich protein 2 (HRP2)/plasmodium lactate dehydrogenase (pLDH) Combo, DiaSys, UK)

SECONDARY OUTCOMES:
Incidence of malaria cases in children 6 months to 10 years | Two years post intervention follow up
  Malaria incidence cases will be assessed using Malaria Rapid Diagnostic test (CareStart)
Prevalence of anaemia in children under 5 years old | 12, 18, 24, 30, 36 months post intervention
  Hemoglobin (Hb) concentration will be tested to assess anaemia (<8 g/dL) using HemoCue Hb 201+.
Indoor Anopheles density | Three years post intervention follow up
  Anopheles density per house per night will be assess every quarter in 8 houses per cluster using light trap. Anopheles density and sporozoite rate will be used to estimate the entomological inoculation rate (EIR)
Sporozoite rate | Three years post intervention follow up
  A sub-samples of Anopheles collected indoor will be tested for Plasmodium falciparum circumsporozoite protein using an ELISA test. Sporozoite rate will be used to estimate the EIR with Anopheles density.
Insecticide content in Long Lasting Insecticidal Net (LLIN) | at 0, 12, 24, 30, 36 months post intervention
  30 LLINs will be collected at yearly interval and Insecticide content in g/kg assessed with High-performance liquid chromatography (HPLC)
Mortality in Anopheles after one hour exposure to every study LLIN | at 0, 6, 12, 18, 24, 30, 36 months post intervention
  30 LLINs will be sampled every 6 months and tested in cone bio assay or tunnel test using resistant Anopheles and susceptible Kisumu Anopheles to assess for bio efficacy. 24, 48 and 72 hours mortality post exposure will be recorded.
LLIN usage | at 6, 12, 18, 24, 30, 36 months post intervention
  The proportion of study participant declaring sleeping under a LLIN the previous night will be assessed during household survey every 6 months using a questionnaire.
Malaria infection prevalence in children 6 months to 14 years | 12 months post intervention
  Malaria prevalence will be assessed using Malaria Rapid Diagnostic test (CareStart Malaria histidine-rich protein 2 (HRP2)/plasmodium lactate dehydrogenase (pLDH) Combo, DiaSys, UK)
Malaria infection prevalence in children 6 months to 14 years | 18 months post intervention
  Malaria prevalence will be assessed using Malaria Rapid Diagnostic test (CareStart Malaria histidine-rich protein 2 (HRP2)/plasmodium lactate dehydrogenase (pLDH) Combo, DiaSys, UK)
Malaria infection prevalence in children 6 months to 14 years | 30 months post intervention
  Malaria prevalence will be assessed using Malaria Rapid Diagnostic test (CareStart Malaria histidine-rich protein 2 (HRP2)/plasmodium lactate dehydrogenase (pLDH) Combo, DiaSys, UK)
Malaria infection prevalence in children 6 months to 14 years | 36 months post intervention
  Malaria prevalence will be assessed using Malaria Rapid Diagnostic test (CareStart Malaria histidine-rich protein 2 (HRP2)/plasmodium lactate dehydrogenase (pLDH) Combo, DiaSys, UK)
Cost & DALYs of each type of bi-treated LLIN | Three years post intervention
  Cost of each intervention will be gathered and used to calculate cost per malaria case averted and cost per DALY averted

OTHER OUTCOMES:
Insecticide resistance intensity in wild Anopheles population | Three years post intervention follow up
  Twice a year insecticide resistance will be assessed in wild Anopheles. 24 hours mortality will be recorded in Anopheles exposed to different concentrations of insecticides in CDC bottle assay or WHO test
P450 over-expression in wild Anopheles population | Three years post intervention follow up
  P450 genes involved in pyrethroid insecticide resistance will be monitored in the 4 arms once a year using reverse-transcription quantitative polymerase chain reaction (PCR)
Frequency of Vgsc mutation in wild Anopheles population | Three years post intervention follow up
  A sub sample of mosquitoes collected in the 4 arms will be tested for the Vgsc mutation involved in pyrethroid resistance using Taq Man PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Natacha Protopopoff, Phd, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- District Misungwi, Misungwi, Mwanza Region, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in each publication will be shared and accessible in the LSHTM repository.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: June 2023
Access Criteria: Upon request

REFERENCES:
- [Background] Mosha JF, Kulkarni MA, Messenger LA, Rowland M, Matowo N, Pitt C, Lukole E, Taljaard M, Thickstun C, Manjurano A, Mosha FW, Kleinschmidt I, Protopopoff N. Protocol for a four parallel-arm, single-blind, cluster-randomised trial to assess the effectiveness of three types of dual active ingredient treated nets compared to pyrethroid-only long-lasting insecticidal nets to prevent malaria transmitted by pyrethroid insecticide-resistant vector mosquitoes in Tanzania. BMJ Open. 2021 Mar 8;11(3):e046664. doi: 10.1136/bmjopen-2020-046664. PMID 34006037
- [Background] Ranson H, N'guessan R, Lines J, Moiroux N, Nkuni Z, Corbel V. Pyrethroid resistance in African anopheline mosquitoes: what are the implications for malaria control? Trends Parasitol. 2011 Feb;27(2):91-8. doi: 10.1016/j.pt.2010.08.004. Epub 2010 Sep 16. PMID 20843745
- [Background] Asidi A, N'Guessan R, Akogbeto M, Curtis C, Rowland M. Loss of household protection from use of insecticide-treated nets against pyrethroid-resistant mosquitoes, benin. Emerg Infect Dis. 2012 Jul;18(7):1101-6. doi: 10.3201/eid1807.120218. PMID 22709930
- [Background] Ochomo EO, Bayoh NM, Walker ED, Abongo BO, Ombok MO, Ouma C, Githeko AK, Vulule J, Yan G, Gimnig JE. The efficacy of long-lasting nets with declining physical integrity may be compromised in areas with high levels of pyrethroid resistance. Malar J. 2013 Oct 24;12:368. doi: 10.1186/1475-2875-12-368. PMID 24156715
- [Result] Mosha JF, Kulkarni MA, Lukole E, Matowo NS, Pitt C, Messenger LA, Mallya E, Jumanne M, Aziz T, Kaaya R, Shirima BA, Isaya G, Taljaard M, Martin J, Hashim R, Thickstun C, Manjurano A, Kleinschmidt I, Mosha FW, Rowland M, Protopopoff N. Effectiveness and cost-effectiveness against malaria of three types of dual-active-ingredient long-lasting insecticidal nets (LLINs) compared with pyrethroid-only LLINs in Tanzania: a four-arm, cluster-randomised trial. Lancet. 2022 Mar 26;399(10331):1227-1241. doi: 10.1016/S0140-6736(21)02499-5. PMID 35339225
- [Derived] Lukole EA, Cook J, Mosha JF, Matowo NS, Kulkarni MA, Mallya E, Aziz T, Martin J, Rowland M, Kleinschmidt I, Manjurano A, Mosha FW, Protopopoff N. Community benefits of mass distribution of three types of dual-active-ingredient long-lasting insecticidal nets against malaria prevalence in Tanzania: evidence from a 3-year cluster-randomized controlled trial. BMC Public Health. 2025 Jan 28;25(1):346. doi: 10.1186/s12889-025-21586-x. PMID 39875853
- [Derived] Lukole EA, Cook J, Mosha JF, Mallya E, Aziz T, Kulkarni MA, Matowo NS, Martin J, Rowland M, Kleinschmidt I, Manjurano A, Mosha FW, Protopopoff N. Will a lack of fabric durability be their downfall? Impact of textile durability on the efficacy of three types of dual-active-ingredient long-lasting insecticidal nets: a secondary analysis on malaria prevalence and incidence from a cluster-randomized trial in north-west Tanzania. Malar J. 2024 Jun 28;23(1):199. doi: 10.1186/s12936-024-05020-y. PMID 38943155
- [Derived] Mosha JF, Matowo NS, Kulkarni MA, Messenger LA, Lukole E, Mallya E, Aziz T, Kaaya R, Shirima BA, Isaya G, Taljaard M, Hashim R, Martin J, Manjurano A, Kleinschmidt I, Mosha FW, Rowland M, Protopopoff N. Effectiveness of long-lasting insecticidal nets with pyriproxyfen-pyrethroid, chlorfenapyr-pyrethroid, or piperonyl butoxide-pyrethroid versus pyrethroid only against malaria in Tanzania: final-year results of a four-arm, single-blind, cluster-randomised trial. Lancet Infect Dis. 2024 Jan;24(1):87-97. doi: 10.1016/S1473-3099(23)00420-6. Epub 2023 Sep 27. PMID 37776879
- [Derived] Messenger LA, Matowo NS, Cross CL, Jumanne M, Portwood NM, Martin J, Lukole E, Mallya E, Mosha JF, Kaaya R, Moshi O, Pelloquin B, Fullerton K, Manjurano A, Mosha FW, Walker T, Rowland M, Kulkarni MA, Protopopoff N. Effects of next-generation, dual-active-ingredient, long-lasting insecticidal net deployment on insecticide resistance in malaria vectors in Tanzania: an analysis of a 3-year, cluster-randomised controlled trial. Lancet Planet Health. 2023 Aug;7(8):e673-e683. doi: 10.1016/S2542-5196(23)00137-7. PMID 37558348
- [Derived] Martin JL, Messenger LA, Mosha FW, Lukole E, Mosha JF, Kulkarni M, Churcher TS, Sherrard-Smith E, Manjurano A, Protopopoff N, Rowland M. Durability of three types of dual active ingredient long-lasting insecticidal net compared to a pyrethroid-only LLIN in Tanzania: methodology for a prospective cohort study nested in a cluster randomized controlled trial. Malar J. 2022 Mar 19;21(1):96. doi: 10.1186/s12936-022-04119-4. PMID 35305667